CLINICAL TRIAL: NCT06764615
Title: A Phase 2, Open-Label Extension Trial to Evaluate the Long-term Safety and Tolerability of Oral Zasocitinib (TAK-279) in Participants With Moderately to Severely Active Ulcerative Colitis and Moderately to Severely Active Crohn's Disease
Brief Title: A Continuation Study of TAK-279 in Adults With Ulcerative Colitis (UC) and Crohn's Disease (CD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-279-IBD-2001; 2024-518914-18-00 (EU CTIS Number: EU CTR Number)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crohn's Disease: Zasocitinib (Experimental): Participants with Crohn's Disease (CD) who completed Week 52 of the parent study, TAK-279-CD-2001 (NCT06233461) will be enrolled in this open-label extension trial to receive Zasocitinib, orally, once daily for up to 108 weeks.
  Interventions: Drug: Zasocitinib
- Ulcerative Colitis: Zasocitinib (Experimental): Participants with Ulcerative Colitis (UC) who completed Week 52 of the parent study, TAK-279-UC-2001 (NCT06254950) will be enrolled in this open-label extension trial to receive Zasocitinib, orally, once daily for up to 108 weeks.
  Interventions: Drug: Zasocitinib

INTERVENTIONS:
Drug: Zasocitinib — Zasocitinib capsules.
  Other Names: TAK-279

SUMMARY:
Crohn's Disease and Ulcerative Colitis are two types of inflammatory bowel disease (IBD), which is a serious, long-term condition in the gut (intestine) that can cause pain and swelling (inflammation) in the bowel. TAK-279 is a medicine which helps to block inflammation.

This study is an extension of the parent studies, TAK-279-CD-2001 (NCT06233461) and TAK-279-UC-2001 (NCT06254950). This means that participants who responded to treatment with TAK-279 in either of the parent studies may be able to continue to benefit from the treatment in this study.

The main aim of this study is to find out how safe TAK-279 is for long term use and to check if it reduces bowel inflammation and symptoms when used for a longer period of time in adults with moderately to severely active UC or CD.

The participants will be treated with TAK-279 for up to 2 years (108 weeks).

During the study, participants will visit their study clinic 11 times.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing and able to understand and fully comply with trial procedures and requirements (including digital tools and applications), in the opinion of the investigator.

   The participant has provided informed consent (that is, in writing, documented via a signed and dated informed consent form [ICF]) and any required privacy authorization prior to the initiation of any trial procedures.

   Disease-Specific Inclusion Criteria:
2. Completion of Week 52 in the parent phase 2 CD and UC trials with valid electronic (e) Diary data for Week 52 (TAK-279-CD-2001 and TAK-279-UC-2001).
3. Clinical or symptomatic responder at parent trial Week 52 as defined below:

   1. TAK-279-CD-2001: Clinical response in PRO2 at parent trial Week 52, assessed as >=30% decrease in average daily very soft or liquid stools and/ or >=30% decrease in average AP from parent trial baseline.
   2. TAK-279-UC-2001: Symptomatic response at parent trial Week 52, assessed as a reduction in partial modified Mayo score (pmMS) of >=1 points and >=30% from parent trial baseline; and a decrease from parent trial baseline in the rectal bleeding sub-score of >=1 point or an absolute rectal bleeding sub-score of <=1 point.

   Other General Inclusion Criteria:
4. Participants must meet the contraception recommendations.

Exclusion Criteria:

1. Participant considered by the investigator to be unsuitable for the OLE trial due to their trial compliance and medication adherence concerns.
2. Participants with malignancy or dysplasia per endoscopy any time during the parent trial or at the beginning of the OLE.

   Exclusion Criteria related to Laboratory Investigations:
3. Participants meeting the exclusion criteria related to laboratory investigations as defined in the protocol.

   Exclusion criteria related to other prohibited concomitant medication:
4. Participants taking oral corticosteroids for CD or UC during parent trial at or after Week 48.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESIs) | From start of study drug administration up to Week 112 (current study)
  TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product. An AESI is an adverse event of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator may be appropriate.
Number of Participants With Clinically Significant Changes in Vital Sign Values | From start of study drug administration up to Week 112 (current study)
  Vital sign values include body temperature, respiratory rate, sitting blood pressure (systolic and diastolic, resting more than 5 minutes), pulse (beats per minute). Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in Clinical Laboratory Values | From start of study drug administration up to Week 112 (current study)
  Laboratory parameters include hematology, clinical chemistry and urinalysis. Clinical significance of laboratory values will be determined at the investigator's discretion.
Number of Participants With Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Values | At Day 1 and Week 108 (current study)
  ECGs will be performed with the participant in the supine or semi-supine position and after resting comfortably for at least 5 minutes. Clinical significance of 12-lead ECG values will be determined at the investigator's discretion.

SECONDARY OUTCOMES:
Percentage of CD Participants Achieving Clinical Remission Based on the Crohn's Disease Activity Index (CDAI) | Up to Week 108 (current study)
  Clinical remission is defined as a CDAI score of less than (<) 150 points.
Percentage of CD Participants Achieving Clinical Response Based on the CDAI | Up to Week 108 (current study)
  Clinical response is defined as greater than (>) 100-point decrease from parent study baseline in CDAI score.
Percentage of CD Participants Achieving Decrease in Endoscopic Response Based on Simple Endoscopic Score for Crohn's Disease (SES-CD) | At Weeks 48 and 108 (current study)
  Endoscopic response is defined by decrease in SES-CD >50 percent (%) from baseline (defined as baseline in parent study TAK-279-CD-2001 [NCT06233461]) (or for participants with isolated ileal disease, SES-CD less than (<) 4 or at least a 2-point reduction from baseline). The SES-CD score ranges from 0 to 56 which includes 4 endoscopic variables (intestinal surface affected by ulcers, intestinal surface affected by other inflammatory lesions, presence of ulcers, and presence of narrowing).
Percentage of CD Participants Achieving Endoscopic Remission Based on SES-CD | At Weeks 48 and 108 (current study)
  Endoscopic remission is defined as SES-CD score <4 or <2 for ileal disease, no sub-score >1. The SES-CD score ranges from 0 to 56 which includes 4 endoscopic variables (the intestinal surface affected by ulcers, the intestinal surface affected by other inflammatory lesions, the presence of ulcers, and the presence of narrowing).
Percentage of CD Participants With Clinical Remission in 2-item Patient-reported Outcome Measure (PRO2) | Up to Week 108 (current study)
  Clinical remission based on PRO2 is defined as average daily liquid or very soft stool frequency (SF) score less than or equal to (<=) 2.8 and not worse than parent study baseline and average daily abdominal pain (AP) score <=1 and not worse than baseline.
Percentage of CD Participants With a Clinical Response in PRO2 | Up to Week 108 (current study)
  Clinical response based on PRO2 is defined as greater than or equal to (>=) 30% decrease in average daily very soft or liquid stools and/ or >=30% decrease in average AP from parent study baseline.
Percentage of UC Participants Achieving Clinical Remission Based on Modified Mayo Score (mMS) | At Weeks 48 and 108 (current study)
  The mMS is a composite score of 3 assessments consisting of stool frequency (SF), rectal bleeding (RB), and endoscopic score (ES). Each component sub-score ranges from 0 to 3 and total score range of the mMS is from 0 to 9, with higher scores indicating more severe disease. Clinical remission is defined as Mayo RB sub-score of 0, Mayo SF sub-score of 0 or 1, and ES sub-score 1 or 0 (score of 1 modified to exclude friability).
Percentage of UC Participants Achieving Clinical Response Based on mMS | At Weeks 48 and 108 (current study)
  Clinical response is defined as reduction from parent study baseline in mMS of >=2 points and >=30% from parent study baseline and a decrease from parent study baseline in the RB sub-score of >=1 point or an absolute RB sub-score of <=1 point.
Percentage of UC Participants Achieving a Symptomatic Remission | Up to Week 108 (current study)
  Symptomatic remission is defined as RB sub-score of 0 and SF sub-score of Mayo score <=1.
Percentage of UC Participants Achieving Endoscopic Improvement Based on Modified Mayo Endoscopic Sub-score (ES) | At Weeks 48 and 108 (current study)
  Endoscopic improvement is defined as a modified Mayo ES of <=1 (score of 1 modified to exclude friability).
Percentage of UC Participants Achieving Endoscopic Remission Based on Modified Mayo (ES) | At Weeks 48 and 108 (current study)
  Endoscopic remission is defined as a modified Mayo ES of 0.
Percentage of CD or UC Participants With no Bowel Urgency | Up to Week 108 (current study)
  Bowel urgency is measured by the bowel urgency electronic diary (eDiary) item.
Percentage of UC or CD Participants With no Abdominal Pain | Up to Week 108 (current study)
  Abdominal pain is measured by abdominal pain eDiary item.
Change From Baseline in Fatigue in UC or CD Participants as Measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score | Up to Week 108 (current study)
  The FACIT-Fatigue is a reliable and valid instrument for measuring fatigue. The responses to the 13 items on the FACIT-Fatigue questionnaire are each measured on a 5-point Likert scale, where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit and 4=Very much. The total score ranges from 0 to 52. High scores represent less fatigue.
Percentage of UC or CD Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score >=170 | Up to Week 108 (current study)
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel systems (10 items), emotional function (12 items), systemic function (5 items), and social function (5 items). The total score ranges from 32 to 224, with higher scores representing better quality of life.
Change From Baseline in Disease-Specific Health-related Quality of Life (HRQoL) in UC or CD Participants as Measured by IBDQ Total Score | Up to Week 108 (current study)
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel systems (10 items), emotional functional (12 items), systemic function (5 items), and social function (5 items). The total score ranges from 32 to 224, with higher scores representing better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (16):
- United States (2):
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Tyler Research Institute, LLC, Tyler, Texas
- China (4):
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangdong, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
- Hepato-Gastroenterologie HK s.r.o., Hradec Králové, Czechia
- Pannonia Maganorvosi Centrum, Budapest, Hungary
- St. Antonius Ziekenhuis, Tilburg, North Brabant, Netherlands
- Poland (4):
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne MedykSp. z o.o. Sp. K., Lublin
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Endomed, Košice, Slovakia
- South Korea (2):
  - Inje University Haeundae Paik Hospital, Haeundae, Busan Gwangyeogsi
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/3da1ed30e4714bf0??page=1&idFilter=TAK-279-IBD-2001